CLINICAL TRIAL: NCT07399951
Title: WU 409: Immune Responses to Rabies Vaccine in the Presence and Absence of Neutralizing Antibodies
Brief Title: Washington University WU 409: Immune Responses to Rabies Vaccine.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Rachel Presti, Professor in Department of Medicine, Division of Infectious Disease Washington University, St. Louis, MO, Washington University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202305094; PJ000006488 (Other Grant/Funding Number: Institutional Grant/Award Human Clinical Studies fund)
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2023-07

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: RANDOMIZATION PROCEDURES Participants will be randomized 1:1 to either:
  Arm-1 Imovax or RabAvert- 2 doses 7 days apart or Arm 2 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 0 Once 5 participants are enrolled to arms 1 and 2 participants will be randomized 1:3 to either Arm-1 Imovax or RabAvert- 2 doses 7 days apart or Arm 2 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 0 Arm 3 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 28
  TO
  RANDOMIZATION PROCEDURES Participants will be randomized 1:1 to either:
  Arm-1 Imovax or RabAvert- 2 doses 7 days apart or Arm-2 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 0
  Once 20 participants are enrolled to arms 1 and 2 10 more participants will be enrolled to:
  Arm-3 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 28
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm-1 Imovax or RabAvert- 2 doses 7 days apart (Experimental): Imovax or RabAvert- 2 doses 7 days apart
  Interventions: Drug: Imovax; Drug: RabAvert
- Arm 2 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 0 (Experimental): Imovax or RabAvert- 2 doses 7 days apart with RIG at day 0
  Interventions: Drug: Imovax; Drug: RabAvert; Drug: HyperRAB
- Arm 3 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 28 (Experimental): Imovax or RabAvert- 2 doses 7 days apart with RIG at day 28
  Interventions: Drug: Imovax; Drug: RabAvert; Drug: HyperRAB

INTERVENTIONS:
Drug: Imovax — Rabies Vaccine
Drug: RabAvert — Rabies Vaccine
  Other Names: RabAver
Drug: HyperRAB — rabies immune globulin (human)
  Arms: Arm 2 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 0; Arm 3 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 28

SUMMARY:
This study will evaluate the immune response to rabies vaccination persons 18 years and older. We will evaluate thirty healthy participants across three cohorts: 1) standard rabies pre-exposure prophylaxis regimen (two doses of Imovax® or RabAvert® seven days apart with no RIG); 2) rabies pre-exposure prophylaxis regimen + day 0 RIG (two doses of Imovax® or RabAvert® seven days apart, with RIG administered at day 0); 3) rabies pre-exposure prophylaxis regimen + day 28 RIG (two doses of Imovax® or RabAvert® seven days apart, with RIG administered at day 28).

DETAILED DESCRIPTION:
This study will evaluate the immune response to rabies vaccination persons 18 years and older. We will evaluate thirty healthy participants across three cohorts: 1) standard rabies pre-exposure prophylaxis regimen (two doses of Imovax® or RabAvert® seven days apart with no RIG); 2) rabies pre-exposure prophylaxis regimen + day 0 RIG (two doses of Imovax® or RabAvert® seven days apart, with RIG administered at day 0); 3) rabies pre-exposure prophylaxis regimen + day 28 RIG (two doses of Imovax® or RabAvert® seven days apart, with RIG administered at day 28).

RANDOMIZATION PROCEDURES Participants will be randomized 1:1 to either:

Arm-1 Imovax or RabAvert- 2 doses 7 days apart or Arm-2 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 0

Once 20 participants are enrolled to arms 1 and 2 10 more participants will be enrolled to:

Arm-3 Imovax or RabAvert- 2 doses 7 days apart with RIG at day 28

We plan to enroll 30 evaluable participants in the coming year, anticipating up to 30 enrolling in the optional FNA and BMA assessments

ELIGIBILITY:
Inclusion Criteria:

- 1. Healthy participants over 18 years of age. 2. Able to understand and give informed consent. 3. Willing to receive rabies vaccine 4. In stable health, as determined by medical history and targeted physical exam related to this history.

5. For those willing to give FNA, CBL and BMA samples, Willing to: give FNA specimens OR give CBL specimens OR give bone marrow aspirates OR give both FNA and BMA specimens OR give both FNA and CBL specimens OR give FNA, CBL and BMA specimens

Exclusion Criteria:

1. Receipt of prior rabies vaccination or risk for rabies exposure requiring standard vaccination
2. Has a current or previous diagnosis of immunocompromising condition to include human immunodeficiency virus, immune-mediated disease requiring immunosuppressive treatment, or other immunosuppressive condition.
3. Has received systemic immunosuppressants or immune-modifying drugs for > 14 days in total within 6 months prior to Screening (for corticosteroids ≥ 10 mg/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
4. Is acutely ill or febrile (temperature >38.0 C [100.4F] less than 72 hours prior to or at the day 1 visit. Participants who meet this criteria may be rescheduled.
5. Currently has symptomatic acute or unstable chronic disease requiring medical or surgical care, to include significant change in therapy or hospitalization, at the discretion of the investigator.
6. History of excessive alcohol consumption, drug abuse, psychiatric conditions, social conditions or occupational conditions that in the opinion of the investigator would preclude compliance with the study.
7. Has received any vaccine ≤ 28 days prior to the injection (Day 1) or plans to receive a vaccine within 28 days before or after the study injection. These participants may be rescheduled.
8. Pregnant women and nursing mothers or women who are planning to become pregnant for the study duration.
9. Have donated blood, blood products or bone marrow within 30 days before study vaccination, plan to donate blood at any time during the duration of participant study participation, or plan to donate blood within 30 days after the last blood draw.
10. Any condition in the opinion of the investigator that would interfere with the proper conduct of the trial.
11. Coagulopathy (primary or iatrogenic) which would contraindicate bone marrow aspirate or core lymph node biopsy for participants willing to have those procedures done
12. Known IgA deficiency, as this is a known risk factor for anaphylactic reactions to Rabies immunoglobulin.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison of antibody titers at D28 versus baseline | 28 days
  Comparison of antibody titers at D28 versus baseline
Comparison of antibody titers at D365 versus baseline | 365 days
  Comparison of antibody titers at D365 versus baseline

SECONDARY OUTCOMES:
Frequency serious adverse events | time of consent to day 365
  Number of serious adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Presti, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine Infectious Disease Clinical Trials Unit., St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: ICF is attached Protocol is attached CSR within 30 days of completion.
Access Criteria: ICF is attached Protocol is attached